CLINICAL TRIAL: NCT04047784
Title: Pilot Study to Evaluate the Role of Endobronchial Ultrasound (EBUS) in the Diagnosis of Acute Pulmonary Embolism in Critically Ill Patients
Brief Title: Pilot Study to Evaluate the Role of EBUS in the Diagnosis of Acute PE in Critically Ill Patients
Acronym: VEBUS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Colleen Channick, MD, Clinical Professor of Medicine, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB# 19-000295
Record Dates: First submitted 2019-05-31; First posted 2019-08-07 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Acute Pulmonary Embolism
Keywords: EBUS; Acute Pulmonary Embolism; Endobronchial Ultrasound; Pilot

STUDY DESIGN:
Intervention Model Description: This is a single center, pilot study to evaluate critically ill patients diagnosed with acute pulmonary embolism using endobronchial ultrasound (EBUS). The investigators anticipate to enroll 60 subjects at Ronald Reagan UCLA Medical Center and UCLA Medical Center, Santa Monica. The enrolled subjects will be imaged using the flexible bronchoscopy with EBUS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Critically Ill Patients (Experimental): Intubated patients in the intensive care unit (ICU) where there is a clinical concern for acute pulmonary embolism or a confirmed diagnosis for acute pulmonary embolism.
  The enrolled subjects will be imaged using the flexible bronchoscopy with EBUS.
  Interventions: Device: Endobronchial ultrasound (EBUS)
- Patients undergoing standard of care clinical bronchoscopy (Experimental): Patients undergoing clinical bronchoscopy as a part of their standard of care.
  The enrolled subjects will be imaged using the flexible bronchoscopy with EBUS.
  Interventions: Device: Endobronchial ultrasound (EBUS)
- Previously recorded patient media from standard of care clinical bronchoscopy with EBUS (No Intervention): Patients who underwent a standard of care clinical bronchoscopy with EBUS previously.
  Information and media including images and videos that were previously recorded for patients who underwent a standard of care clinical bronchoscopy with EBUS will be available to the study team.

INTERVENTIONS:
Device: Endobronchial ultrasound (EBUS) — An Olympus EBUS bronchoscope will be used for all endobronchial ultrasound examinations. This scope has a 6.9 mm outer diameter, a 2.7 mm working channel and 30-degree oblique forward-viewing optics. A 12 MHz linear ultrasound transducer with a maximum penetration of 50 mm will be linked to a processor (Olympus EU-ME2) that allows an integrated power Doppler mode to visualize the vascular blood flow.
  Bronchoscopy will be introduced through the adaptor connected to the endotracheal tube, in patients who are already under general anesthesia and on mechanical ventilation. The bronchoscope will be advanced into the airways and endobronchial ultrasound of the main pulmonary artery (PA) and lobar branches will be performed in a standardized fashion. At the completion of the imaging the EBUS bronchoscope will be withdrawn.
  Arms: Critically Ill Patients; Patients undergoing standard of care clinical bronchoscopy

SUMMARY:
Acute pulmonary embolism (PE) in critically ill patients is common and often life threatening. The diagnosis of acute PE is often entertained in intensive care unit patients who develop unexplained hypotension or hypoxemia. Obtaining diagnostic confirmation of acute PE with a contrast-enhanced computed tomography of the chest (CT angiogram) may be difficult as patients are often too unstable for transport to the CT scanner or have renal insufficiency limiting the ability to receive intravenous contrast agents. Making or excluding the diagnosis of acute PE in these patients is critically important, as hemodynamic instability or right heart dysfunction, if due to PE, puts patients in the massive or submassive category and increased mortality risk. More aggressive therapies such as thrombolysis, extracorporeal membrane oxygenation or surgical embolectomy are often entertained. The investigators have previously described a case where endobronchial ultrasound (EBUS) was employed in the diagnostic algorithm of suspected acute PE and significantly affected treatment recommendations. The investigators believe that, in these patients, use of EBUS to assess for thrombotic occlusion of the central pulmonary vasculature can fill a critical gap in the decision tree for management of these patients.

EBUS has become part of the diagnostic approach in a number of clinical situations, including the workup and staging of suspected malignancy, unexplained lymphadenopathy, and diagnosis of mediastinal and parabronchial masses. There is strong evidence that EBUS is equivalent to mediastinoscopy in the mediastinal staging of lung cancer. The number of physicians skilled and experienced in performance of EBUS has increased dramatically, and training in the procedure is frequently obtained in a pulmonary fellowship.

To our knowledge, there have been no prospective studies that investigate the use of EBUS as a tool for the diagnosis of acute central pulmonary embolism in critically ill patients where obtaining diagnostic confirmation of this diagnosis with a contrast-enhanced computed tomography of the chest is not safe or feasible.

DETAILED DESCRIPTION:
This is a single center, pilot study to evaluate critically ill patients diagnosed with acute pulmonary embolism using endobronchial ultrasound (EBUS). The investigators anticipate to enroll 20 subjects at Ronald Reagan UCLA Medical Center and UCLA Medical Center, Santa Monica. The enrolled subjects will be imaged using the flexible bronchoscopy with EBUS.

After informed consent is obtained, the following procedure will be performed:

An Olympus EBUS bronchoscope will be used for all endobronchial ultrasound examinations. This scope has a 6.9 mm outer diameter, a 2.7 mm working channel and 30-degree oblique forward-viewing optics. A 12 MHz linear ultrasound transducer with a maximum penetration of 50 mm will be linked to a processor (Olympus EU-ME2) that allows an integrated power Doppler mode to visualize the vascular blood flow.

Bronchoscopy will be introduced through the adaptor connected to the endotracheal tube, in patients who are already under general anesthesia and on mechanical ventilation. The bronchoscope will be advanced into the airways and endobronchial ultrasound of the main pulmonary artery (PA) and lobar branches will be performed in a standardized fashion as follow:

Advance the bronchoscopy into the right main bronchus distally to the level of the right lower lobe, between 12 and 3 o'clock position where the interlobar artery of the PA is seen. Then the scope will be pulled back slowly, turning counterclockwise, following the course of the PA on the medial wall of the right bronchial tree until the level of the carina, where the right main PA and the PA trunk are seen. The scope is then turned to the right again, towards 3 o'clock following the right upper lobe bronchus to examine the upper lobar artery. The scope is then advanced into the left main bronchus, towards 9 o'clock to examine the upper lobar artery, then advanced distally to the left lower lobe bronchus to examine the interlobar artery. At the completion of the imaging the EBUS bronchoscope will be withdrawn.

Ultrasound images and video will be stored to the machine and visualized thrombi will be marked.

For patients who have had a chest CT for suspected PE, the investigators will assess sensitivity and specificity of EBUS to visualize or exclude PE. For patients who are unable to have a CT, the investigators will not be able to determine true efficacy, but will report the number of positive and negative studies and follow these patients for outcome and subsequent definitive diagnosis of venous thromboembolism.

As this is a pilot study looking at the feasibility of EBUS for diagnosing acute pulmonary embolism, study personnel performing the EBUS will not be blinded to the clinical diagnosis and the management of the subject. A brief report of the procedure results will be uploaded in the patient's medical record. Any clinically relevant findings from the EBUS will be communicated to the subject's treating team. Regardless of the findings, a note stating that the EBUS technique is not yet established for evaluating acute pulmonary embolism in critically ill patients will be emphasized in order to prevent any bias in the patient's clinical care.

Pulmonary Vascular Mapping Substudy:

Of the 60 total subjects enrolled in the study, approximately 20 subjects under the criteria below will be enrolled at Ronald Reagan UCLA Medical Center and UCLA Medical Center, Santa Monica undergoing clinical bronchoscopy as a part of their standard of care. The enrolled subjects will be imaged using the flexible bronchoscopy with EBUS.

Retrospective Chart Review:

Of the 60 total subjects enrolled in the study, media including images and videos that are previously recorded for 20 patients who underwent a clinical bronchoscopy with EBUS as a part of their standard of care will also be available to our research team without consent from the patient to help supplement the data we obtain from the 20 subjects that are enrolled in the pulmonary vascular mapping substudy.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age.
* The patient or patient's surrogate must understand and sign informed consent form (ICF).
* Intubated patients in the intensive care unit (ICU) where there is a clinical concern for acute pulmonary embolism or a confirmed diagnosis for acute pulmonary embolism.

Exclusion Criteria:

* Patient does not meet the requirements to undergo clinical bronchoscopy, as determined by the treating physician.
* Endotracheal tube size less than 8.0 mm.
* Contraindications to lidocaine.

Pulmonary Vascular Mapping Substudy:

Enrollment for the pulmonary vascular mapping substudy will be based on the following inclusion and exclusion criteria:

Inclusion criteria:

* Patient ≥ 18 years of age.
* The patient or patient's surrogate must understand and sign informed consent form (ICF).
* Intubated patients undergoing clinical bronchoscopy, as determined by the treating physician.

Exclusion criteria:

* Patient does not meet the requirements to undergo clinical bronchoscopy, as determined by the treating physician.
* Endotracheal tube size less than 8.0 mm.
* Contraindications to lidocaine.

Retrospective Chart Review:

Of the 60 total subjects enrolled in the study, media including images and videos that are previously recorded for 20 patients who underwent a clinical bronchoscopy with EBUS as a part of their standard of care will also be available to our research team without consent from the patient to help supplement the data we obtain from the 20 subjects that are enrolled in the pulmonary vascular mapping substudy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-08-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CT angiogram results (if obtained) | 2 years
  For patients who have had a chest CT for suspected PE, the investigators will obtain a copy of the participant's chest CT for suspected PE report.
Patient treatment | 2 years
  For patients who are unable to have a CT, the investigators will not be able to determine true efficacy, but will report the number of positive and negative studies. Patient treatment will be reported as:
  * Catheter Directed Lysis
  * Heparin Drip
  * Surgical Embolectomy
  * Thrombolysis
  * No Treatment for Pulmonary Embolism (PE)
Patient outcome | 2 years
  For patients who are unable to have a CT, the investigators will not be able to determine true efficacy, but follow these patients for outcome and subsequent definitive diagnosis of venous thromboembolism. Subsequent patient outcome will be reported as:
  * Alive
  * Extended hospitalization
  * Intervention to prevent impairment or damage
  * Life-threatening condition
  * Disability
  * Death
Assess sensitivity and specificity of EBUS to visualize or exclude PE compared to the chest CT. | 2 years
  Ability for EBUS will be reported by its ability to identify each major branch and reporting what branched not identified as:
  * Main Pulmonary Artery (MPA)
  * Right Pulmonary Artery (RPA)
  * Truncus Anterior (TA) or Ascending Branch
  * Right Interlobar Artery or Descending Branch
  * Right Basal Trunk
  * Left Pulmonary Artery (LPA)
  * Left Interlobar Artery
  * Left Basal Trunk
  * Other
Report any complications | 2 years
  Complications during or after the procedure will be reported as:
  * Airway Bleeding
  * Airway Injury
  * Hypotension as defined by < 65 mmHg or need to escalate vasopressors
  * Hypoxia as defined by < 90%
  * Other
  * None
Assess sensitivity and specificity of EBUS to visualize or exclude PE by its ability to identify a clot. | 2 years
  Ability for EBUS will be reported by its ability to identify a clot and reporting the location of the clot as:
  * Main Pulmonary Artery (MPA)
  * Right Pulmonary Artery (RPA)
  * Truncus Anterior (TA) or Ascending Branch
  * Right Interlobar Artery or Descending Branch
  * Right Basal Trunk
  * Left Pulmonary Artery (LPA)
  * Left Interlobar Artery
  * Left Basal Trunk
  * Other
Assess sensitivity and specificity of EBUS to visualize or exclude PE by its ability to identify flow around clot(s) present. | 2 years
  Ability for EBUS will be reported by its ability to identify flow around clot(s) present and reporting the location of the flow around clot(s) present as:
  * Main Pulmonary Artery (MPA)
  * Right Pulmonary Artery (RPA)
  * Truncus Anterior (TA) or Ascending Branch
  * Right Interlobar Artery or Descending Branch
  * Right Basal Trunk
  * Left Pulmonary Artery (LPA)
  * Left Interlobar Artery
  * Left Basal Trunk
  * Other

SECONDARY OUTCOMES:
Other airway finding(s) | 2 years
  Other airway finding(s) will be reported as:
  * Mucus
  * Blood
  * Other

CONTACTS AND LOCATIONS:
Overall Officials: Colleen L Channick, M.D., Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Medical Center, Santa Monica, Santa Monica, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tapson VF. Acute pulmonary embolism. N Engl J Med. 2008 Mar 6;358(10):1037-52. doi: 10.1056/NEJMra072753. No abstract available. PMID 18322285
- [Background] Stein PD, Henry JW. Prevalence of acute pulmonary embolism among patients in a general hospital and at autopsy. Chest. 1995 Oct;108(4):978-81. doi: 10.1378/chest.108.4.978. PMID 7555172
- [Background] Aumiller J, Herth FJ, Krasnik M, Eberhardt R. Endobronchial ultrasound for detecting central pulmonary emboli: a pilot study. Respiration. 2009;77(3):298-302. doi: 10.1159/000183197. Epub 2008 Dec 9. PMID 19065053
- [Background] Ernst A, Anantham D, Eberhardt R, Krasnik M, Herth FJ. Diagnosis of mediastinal adenopathy-real-time endobronchial ultrasound guided needle aspiration versus mediastinoscopy. J Thorac Oncol. 2008 Jun;3(6):577-82. doi: 10.1097/JTO.0b013e3181753b5e. PMID 18520794
- [Background] Yasufuku K, Pierre A, Darling G, de Perrot M, Waddell T, Johnston M, da Cunha Santos G, Geddie W, Boerner S, Le LW, Keshavjee S. A prospective controlled trial of endobronchial ultrasound-guided transbronchial needle aspiration compared with mediastinoscopy for mediastinal lymph node staging of lung cancer. J Thorac Cardiovasc Surg. 2011 Dec;142(6):1393-400.e1. doi: 10.1016/j.jtcvs.2011.08.037. Epub 2011 Oct 2. PMID 21963329
- [Background] Tanner NT, Pastis NJ, Silvestri GA. Training for linear endobronchial ultrasound among US pulmonary/critical care fellowships: a survey of fellowship directors. Chest. 2013 Feb 1;143(2):423-428. doi: 10.1378/chest.12-0212. PMID 22878834
- [Background] Torbicki A, Galie N, Covezzoli A, Rossi E, De Rosa M, Goldhaber SZ; ICOPER Study Group. Right heart thrombi in pulmonary embolism: results from the International Cooperative Pulmonary Embolism Registry. J Am Coll Cardiol. 2003 Jun 18;41(12):2245-51. doi: 10.1016/s0735-1097(03)00479-0. PMID 12821255
- See also: Pulmonary Artery Anatomy — https://www.med-ed.virginia.edu/courses/rad/ctpa/02anat/anat-01-01.html